CLINICAL TRIAL: NCT03995693
Title: Fuel Selection During Eccentric Cycling: Comparison With Concentric Cycling and the Effect of Glucose Ingestion During Exercise
Brief Title: Fuel Selection During Eccentric Cycling With Glucose Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Jonathan Tremblay, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: eccentric-exogenous
Record Dates: First submitted 2019-05-24; First posted 2019-06-24 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Exercise; Damage Muscle; Nutrition
Keywords: eccentric exercise; 13C-glucose; exercise mode
MeSH Terms: conditions — Motor Activity | interventions — Blood Specimen Collection; Electromyography

STUDY DESIGN:
Who Masked: Participant
Masking Description: Opaque bottles to administer beverages with similar sweet taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Concentric cycling with placebo ingestion (Experimental): Participants will complete 45 minutes of arm cranking at an intensity corresponding to 30% of the concentric cycling VO2max, followed by 35 minutes of CONCENTRIC cycling on a recumbent ergometer at the same VO2. A PLACEBO solution (water with a non-caloric sweetener) will be ingested 30 min prior to starting exercise and every 15 min thereafter, until the exercise is completed. Indirect respiratory calorimetry, expired gas sampling, blood sampling will occur will be performed 4 minutes before each ingestion.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load arm cranking; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Procedure: Blood sampling; Behavioral: Measure of maximal voluntary contraction force production; Diagnostic Test: Measure of muscle electrical activity (EMG); Diagnostic Test: Measure of central and cutaneous temperatures; Diagnostic Test: Measure of perceived exertion, pain perception and affective response; Procedure: Measure of sweat and urine production
- Concentric cycling with glucose ingestion (Experimental): Participants will complete 45 minutes of arm cranking at an intensity corresponding to 30% of the concentric cycling VO2max, followed by 35 minutes of concentric cycling on a recumbent ergometer at the same VO2. A GLUCOSE solution (glucose with a trace amount of 13C) will be ingested 30 min prior to starting exercise and every 15 min thereafter, until the exercise is completed. Indirect respiratory calorimetry, expired gas sampling, blood sampling will occur will be performed 4 minutes before each ingestion.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load arm cranking; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Procedure: Blood sampling; Behavioral: Measure of maximal voluntary contraction force production; Diagnostic Test: Measure of muscle electrical activity (EMG); Diagnostic Test: Measure of central and cutaneous temperatures; Diagnostic Test: Measure of perceived exertion, pain perception and affective response; Procedure: Measure of sweat and urine production
- Eccentric cycling with placebo ingestion (Experimental): Participants will complete 45 minutes of arm cranking at an intensity corresponding to 30% of the concentric cycling VO2max, followed by 35 minutes of ECCENTRIC cycling on a recumbent ergometer at the same VO2. A PLACEBO solution (water with a non-caloric sweetener) will be ingested 30 min prior to starting exercise and every 15 min thereafter, until the exercise is completed. Indirect respiratory calorimetry, expired gas sampling, blood sampling will occur will be performed 4 minutes before each ingestion.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load arm cranking; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Procedure: Blood sampling; Behavioral: Measure of maximal voluntary contraction force production; Diagnostic Test: Measure of muscle electrical activity (EMG); Diagnostic Test: Measure of central and cutaneous temperatures; Diagnostic Test: Measure of perceived exertion, pain perception and affective response; Procedure: Measure of sweat and urine production
- Eccentric cycling with glucose ingestion (Experimental): Participants will complete 45 minutes of arm cranking at an intensity corresponding to 30% of the concentric cycling VO2max, followed by 35 minutes of ECCENTRIC cycling on a recumbent ergometer at the same VO2. A GLUCOSE solution (glucose with a trace amount of 13C) will be ingested 30 min prior to starting exercise and every 15 min thereafter, until the exercise is completed. Indirect respiratory calorimetry, expired gas sampling, blood sampling will occur will be performed 4 minutes before each ingestion.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load arm cranking; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Procedure: Blood sampling; Behavioral: Measure of maximal voluntary contraction force production; Diagnostic Test: Measure of muscle electrical activity (EMG); Diagnostic Test: Measure of central and cutaneous temperatures; Diagnostic Test: Measure of perceived exertion, pain perception and affective response; Procedure: Measure of sweat and urine production

INTERVENTIONS:
Dietary Supplement: Solution ingestion — Two ingestion modalities will be attributed (participant is blinded) in random order: a placebo and a glucose solution. The placebo contains water and a non-caloric sweetener (stevia) in order to reproduce the taste of the glucose solution. The glucose solution contains 6% glucose per volume, labelled with 13C. Both solutions will be administered in 8 doses: a bolus (333 mL) at rest, 30 minutes before the start of exercise, 167 mL immediately before exercise, 167 mL every 15 minutes during arm cranking, 125 mL immediately before concentric or eccentric pedalling and at 15 and 25 minutes of this last exercise period. In total, 1250 mL of solution will be administered during the experimental protocol.
Behavioral: Constant load arm cranking — The participants will perform 45 minutes of arm cranking on a specialized ergometer at a power output corresponding to 30% of their concentric cycling VO2max, previously measured.
Procedure: Expired gas sampling — Subjects will be asked, twice, to provide a forced expiration into a 10 mL plastic tube in order to collect a sample expired gases. This procedure will be done immediately before blood sampling and ingestion of the solution.
Procedure: Indirect respiratory calorimetry — A mouthpiece and nose plug will be placed on the subject and expired gases will be analyzed by a metabolic cart during 3 minutes. This procedure will be done immediately before expired gas collection, blood sampling and ingestion of the solution.
Procedure: Blood sampling — A catheter will be inserted in an antecubital vein and a saline solution will be continuously perfused to maintain vein open. 10 mL of blood will be collected immediately before ingesting the solution for a total of 80 mL.
Behavioral: Measure of maximal voluntary contraction force production — Maximal voluntary bilateral knee extensions (3 trials of 3-4 seconds each) will be performed on a chair equipped with force sensors to measure peak force production. These measurements will be done before the first ingestion, immediately before exercise, during the transition between arm cranking and concentric or eccentric cycling, and at the end of the exercise protocol.
Diagnostic Test: Measure of muscle electrical activity (EMG) — Surface electrodes will be placed on the biceps and quadriceps to measure EMG throughout the exercise protocol.
Diagnostic Test: Measure of central and cutaneous temperatures — Wireless sensors will be placed on the skin of the arm, chest, back, abdomen, thigh and calf using adhesive tape. A wireless thermometric pill will be ingested the morning of the experiment. These will allow the measurement of skin and central temperatures throughout the exercise protocol.
Diagnostic Test: Measure of perceived exertion, pain perception and affective response — 100 points scales (CR100) will be used to measure perceived exertion and pain perception immediately before ingesting the gas sampling. At the same time, affective responses will be assessed using the "Feeling scale".
Procedure: Measure of sweat and urine production — Sweat production and sampling will be performed by measuring body weight before and after exercise, after voiding the bladder. Mass loss through the urine and gases will be accounted for in order to compute sweat production. A sweat sample will be collected using a cotton gauze placed into a plastic collector affixed in the upper back of the participants. A urine sample will be taken from the urine collected at the end of the exercise period. Urine and sweat volumes along with respective urea concentrations will be used to compute protein oxidation during exercise.

SUMMARY:
This study compares fuel selection during eccentric and concentric cycling, with (placebo) or without glucose ingestion during exercise. After a 2-week familiarization and habituation with the ergometers, subjects will complete four experimental conditions in a randomized order: concentric with placebo, eccentric with placebo, concentric with glucose, eccentric with glucose.

DETAILED DESCRIPTION:
Cycling on a cycle ergometer typically requires repeated concentric muscle contractions to push on the pedals and produce mechanical work. An eccentric cycling ergometer has a motor that rotates the cranks with a predetermined torque, the cyclist needs to resist to the movement of the cranks. This leads to eccentric muscle contractions, the work is thus produced while the muscle is lengthening (negative work). This mode of exercise is known to produce a lower oxygen consumption (energy cost) for the same mechanical power output and also leads to muscle damage which can interfere with fuel selection.

ELIGIBILITY:
Inclusion Criteria:

* Low alcohol consumption (<3 drinks/week)
* Non-smokers
* Not regularly taking medication for a known pathology
* Regularly practices endurance sports (cycling, running, etc.)

Exclusion Criteria:

* Intolerant to glucose (according to WHO standards)
* Musculoskeletal injury or illness affecting exercise performance
* Failure to respect protocol guidelines (diet, exercise prior to experimentation, etc.)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Exogenous glucose oxidation | Average over the 35 minutes of eccentric or concentric exercise
  Measured by indirect respiratory calorimetry combined with tracer techniques.
Maximal voluntary force production | Change between baseline and end of exercise
  Measured using isometric bilateral knee extensions
Central and skin temperature | Average over the 35 minutes of eccentric or concentric exercise
  Measured using a thermometric pill and skin-surface electrodes
Perceived exertion | Average over the 35 minutes of eccentric or concentric exercise
  Measured using a Category Ratio scale on 100 points (CR100), 0 signifies no exertion and 100 being maximal effort.

SECONDARY OUTCOMES:
Blood insulin concentration | For 0 minutes corresponds to the beginning of exercise, at -31, -1, 14, 29, 44, 49, 59 and 69 minutes
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure insulin concentration.
Blood glucose concentration | For 0 minutes corresponds to the beginning of exercise, at -31, -1, 14, 29, 44, 49, 59 and 69 minutes
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure glucose concentration.
Blood free-fatty acid concentration | For 0 minutes corresponds to the beginning of exercise, at -31, -1, 14, 29, 44, 49, 59 and 69 minutes
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure free-fatty acid concentration.
Blood lactate concentration | For 0 minutes corresponds to the beginning of exercise, at -31, -1, 14, 29, 44, 49, 59 and 69 minutes
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure lactate concentration.
Total carbohydrate, fat and protein oxidation | Average over the 35 minutes of eccentric or concentric exercise
  Measured by indirect respiratory calorimetry corrected for urea excretion in sweat and urine
Pain perception: VAS | Average over the 35 minutes of eccentric or concentric exercise
  Visual analogue pain scale of 25 cm, relative distance converted to score on 100 points. Higher values correspond to greater pain sensation.
Affective response | Average over the 35 minutes of eccentric or concentric exercise
  Feeling scale, ranging from -5 to +5, reporting the mood (Hardy & Rejeski, 1989). -5 corresponds to very bad and +5 to very good.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tremblay, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Centre d'éducation physique et sportive de l'Université de Montréal (CEPSUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No